CLINICAL TRIAL: NCT04636385
Title: Assessment of Jumping Gap Dimension at Maxillary Teeth in Addition to Selected Anatomical Landmarks Related to Immediate Implant Placement in the Esthetic Zone: Observational Cone-Beam Computed Tomography (CBCT) Study.
Brief Title: Jumping Gap Dimension at Maxillary Teeth: Cone-Beam Computed Tomography (CBCT) Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzy Nabil Naiem, Principal Investigator, Cairo University
Other Study IDs: 12 Nov 2020 Protocol
Record Dates: First submitted 2020-11-09; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Jumping Gap Dimension at Maxillary Teeth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study no intervention — No intervention

SUMMARY:
To assess the important anatomical structures involved in the treatment planning of immediate implants, particularly the jumping gap distance at the different maxillary teeth in the esthetic zone using CBCT analysis. Additional relevant radiographic aspects are evaluated as well to aid in decision making related to immediate implants.

ELIGIBILITY:
Inclusion Criteria:

* teeth at upper jaw including : incisors, laterals, canines and premolars

Exclusion Criteria:

* teeth having: extensive restorations, crowns, implants
* CBCT scans showing scattering
* teeth showing bone loss around them indicative of periodontal disease

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Egyptian Population (Cairo Residents)
Sampling Method: Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Jumping gap | 1 month
  Estimation of the jumping gap dimension at maxillary anterior and premolar teeth at different apico-coronal levels through CBCT analysis by linear measurements in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Hani El Nahass, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It has not yet been decided between the study participants

REFERENCES:
- [Background] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. J Clin Periodontol. 2005 Jun;32(6):645-52. doi: 10.1111/j.1600-051X.2005.00726.x. PMID 15882225
- [Background] Botticelli D, Berglundh T, Lindhe J. Hard-tissue alterations following immediate implant placement in extraction sites. J Clin Periodontol. 2004 Oct;31(10):820-8. doi: 10.1111/j.1600-051X.2004.00565.x. PMID 15367183
- [Background] Lee SL, Kim HJ, Son MK, Chung CH. Anthropometric analysis of maxillary anterior buccal bone of Korean adults using cone-beam CT. J Adv Prosthodont. 2010 Sep;2(3):92-6. doi: 10.4047/jap.2010.2.3.92. Epub 2010 Sep 30. PMID 21165276